CLINICAL TRIAL: NCT00726687
Title: Phase 1b Study of Indibulin in Combination With Capecitabine in Advanced Solid Tumors
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Alaunos Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IBL1005
Record Dates: First submitted 2008-07-29; First posted 2008-08-01 (Estimated); Last update posted 2012-07-19 (Estimated); Status verified 2012-07

CONDITIONS: Advanced Solid Tumors
Keywords: Cancer; Indibulin; Capecitabine; Xeloda
MeSH Terms: conditions — Neoplasms | interventions — indibulin; Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- single (Experimental): Single arm designed to elicit Maximum Tolerated Dose
  Interventions: Drug: indibulin; Drug: capecitabine

INTERVENTIONS:
Drug: indibulin — indibulin, dose escalation, 400-600 mg taken twice every day
Drug: capecitabine — capecitabine, dose escalation, 875 mg/m2- 1250 mg/m2, taken twice daily for 14 days per 21 day cycle
  Other Names: Xeloda

SUMMARY:
This is a phase 1b study of Indibulin in combination with Capecitabine in advanced solid tumors.

DETAILED DESCRIPTION:
The primary objective of the trial is to determine the maximum tolerated dose (MTD) and optimal dosing schedule of indibulin in combination with capecitabine in subjects diagnosed as having advanced solid tumors.

Secondary objectives include the determination of dose-limiting toxicity (DLT), safety and tolerability, and preliminary activity of this combination. In addition, biological activity of indibulin in combination with capecitabine will be evaluated.

Single arm, open label, Phase Ib, dose-escalation study of indibulin in combination with capecitabine in subjects with advanced histologically confirmed, solid tumors for which no standard therapy exists and for whom treatment with capecitabine is considered medically acceptable.

3 subjects will be treated at each dose level. When DLT occurs in 2 or more of 6 or fewer subjects, MAD has been reached and the dose will be reduced to the previous dosing level, which will be considered the MTD.

ELIGIBILITY:
Inclusion Criteria

1. Subjects with advanced, histologically confirmed solid tumors for whom treatment with capecitabine is considered medically acceptable
2. ≥18 years of age
3. ECOG performance score ≤2 (see Appendix 2)
4. Eligible subjects MUST have at least one measurable lesion as defined by RECIST guidelines (see Appendix 3). Measurable lesions MUST NOT have been in a previously irradiated field or injected with biological agents.
5. Life-expectancy ≥12 weeks
6. No more than 2 prior chemotherapy regimens for metastatic disease
7. Subjects on prophylactic anticoagulation (i.e., low-dose warfarin) are eligible provided the coagulation parameter levels are as follows: prothrombin time (INR of prothrombin time) <1.1× institutional ULN
8. Adequate bone marrow, liver and renal function as assessed by the following laboratory requirements to be conducted <2 weeks prior to Study Day 1:

   * Creatinine ≤1.5 × upper limit of normal (ULN) OR a calculated creatinine clearance ≥1.50 cc/min (See Appendix 6 for calculation method)
   * Total bilirubin ≤1.5×ULN
   * Alanine transaminase (ALT) and aspartate transaminase (AST) ≤2.5×ULN (<5×ULN for patients presenting with liver involvement)
   * White blood cell count ≥3.0×109/L
   * Absolute neutrophil count (ANC) ≥1.5×109/L
   * Platelets ≥100×109/L
   * Hemoglobin ≥10 g/dL
9. Written informed consent in compliance with ZIOPHARM policies and the Institutional Review Board (IRB) having jurisdiction over the site
10. Ability and willingness to undergo multiple venous punctures for serum PK sampling
11. For the second phase of the trial (expanded cohort of 10), only capecitabine-naïve subjects will be included; prior therapy with 5-FU will be allowed
12. Each man and woman of childbearing potential must agree to use a reliable method of contraception during the study and for 3 months following his or her last dose of study drug

Exclusion Criteria

1. New York Heart Association (NYHA) functional class ≥3 or myocardial infarction within 6 months (see Appendix 4)
2. Severe renal impairment (creatinine clearance below 30 mL/min)
3. Known dihydropyrimidine dehydrogenase deficiency (DPD)
4. Any evidence of bleeding diathesis or coagulopathy
5. International normalized ration (INR) >1.5, unless the subject is on full-dose warfarin
6. Subjects on full-dose anticoagulants (e.g., warfarin) are eligible provided that both of the following criteria are met:

   * The subject must have an in-range INR (usually between 2 and 3) on a stable dose of oral anticoagulant or on a stable dose of low molecular-weight heparin
   * The subject must not have any active bleeding or pathological condition that carries a high risk of bleeding (e.g., tumor involving major vessels or known varices)
7. Pregnancy and/or lactation. To be enrolled, each woman of childbearing potential must have a negative pregnancy test, which will be repeated at the end of the study.
8. Uncontrolled systemic infection (documented with microbiological studies)
9. Anticancer chemotherapy or immunotherapy within 4 weeks of study entry or at any time during the study or investigational drug therapy outside of this trial during or within 4 weeks of study entry
10. Mitomycin C or nitrosureas should not be given within 6 weeks of study entry.
11. Radiotherapy within 3 weeks of study entry or at any time during the study. For target lesions that have been radiated within 3 months of study entry, only those lesions with documented progression post radiation will be allowed.
12. Surgery within 4 weeks of start of study drug dosing, excluding tumor biopsy for pharmacodynamic parameters
13. History of an invasive second primary malignancy diagnosed within the previous 3 years except for Stage I endometrial/cervical carcinoma or prostate carcinoma treated surgically, and non-melanoma skin cancer
14. Substance abuse or medical, psychological or social conditions that may interfere with the subject's participation in the study or the evaluation of study results
15. Any condition that is unstable or could jeopardize the safety of the subject and his/her compliance with study protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2008-06; Primary Completion 2013-06 (Estimated); Study Completion 2013-06 (Estimated)

PRIMARY OUTCOMES:
toxicities | 6 months

SECONDARY OUTCOMES:
pharmacokinetics | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Lewis, MD, Study Chair — Alaunos Therapeutics
Locations (3):
- United States (3):
  - Indianapolis, Indiana
  - Las Vegas, Nevada
  - Vancouver, Washington

REFERENCES:
- [Derived] Kapoor S, Srivastava S, Panda D. Indibulin dampens microtubule dynamics and produces synergistic antiproliferative effect with vinblastine in MCF-7 cells: Implications in cancer chemotherapy. Sci Rep. 2018 Aug 17;8(1):12363. doi: 10.1038/s41598-018-30376-y. PMID 30120268